CLINICAL TRIAL: NCT01499706
Title: Phase I Clinical Trial of Telephone-delivered Motivational Interviewing to Reduce Sexual Risk Behavior in HIV-positive Persons 45-plus Years of Age
Brief Title: Telephone-delivered Behavioral Interventions to Reduce Risky Sexual Behavior in HIV-positive Late Middle-age and Older Adults
Acronym: MI
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ohio University College of Osteopathic Medicine (Other)
Responsible Party: Principal Investigator, Travis Lovejoy, Ph.D., M.P.H., Health Psychology Fellow, Ohio University College of Osteopathic Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OUCOM-MI-1
Record Dates: First submitted 2011-12-21; First posted 2011-12-26 (Estimated); Last update posted 2011-12-26 (Estimated); Status verified 2011-12

CONDITIONS: Unsafe Sex
Keywords: Motivational Interviewing; Telephone; HIV; AIDS; Older Adults
MeSH Terms: conditions — Unsafe Sex; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Standard of Care Control (No Intervention): Participants will receive standard sexual risk reduction services available to them through medical and community-based organizations
- 1-session motivational interviewing (Experimental): Participants will receive a single session of motivational interviewing delivered over the telephone
  Interventions: Behavioral: 1-session of telephone-administered motivational interviewing
- 4-session motivational interviewing (Experimental): Participants will receive four weekly sessions of motivational interviewing delivered over the telephone.
  Interventions: Behavioral: 4-session telephone-administered motivational interviewing

INTERVENTIONS:
Behavioral: 1-session of telephone-administered motivational interviewing — Participants will receive a single session of telephone-delivered motivational interviewing to reduce sexual risk behavior.
  Arms: 1-session motivational interviewing
Behavioral: 4-session telephone-administered motivational interviewing — Participants will receive four weekly sessions of telephone-delivered motivational interviewing to reduce sexual risk behavior.
  Arms: 4-session motivational interviewing

SUMMARY:
The number of late middle-age and older adults living with HIV/AIDS in the U.S. continues to rise due largely to

* better clinical care and the improved efficacy of highly active antiretroviral therapy that has extended the lives of many HIV-positive persons
* an increase in the number of new HIV infections in older persons. This study tested the efficacy of 1- and 4-session telephone-administered behavioral sexual risk reduction interventions for HIV-positive adults 45-plus years of age who engage in risky sexual behaviors.

DETAILED DESCRIPTION:
The number of late middle-age and older adults living with HIV/AIDS in the U.S. continues to rise. In fact, it is estimated that by 2014, 50% of all HIV-positive persons will be 50 years of age or older, due largely to a) better clinical care and the improved efficacy of highly active antiretroviral therapy that has extended the lives of many HIV-positive persons and b) an increase in the number of new HIV infections in older persons. Despite escalating HIV incidence and prevalence rates in older adults, and the fact that an estimated 13% to 30% of older persons living with HIV/AIDS continue to engage in risky sexual practices, few secondary risk reduction interventions have been contextualized to meet the unique needs of sexually active HIV-infected older adults. These unique needs include biological and libidinal changes associated with aging such as erectile dysfunction and the increased use of erectile dysfunction medications in older men, sexual partnerships with younger persons, survivor guilt over outliving romantic partners, and the impact of co-morbid chronic illnesses (e.g., diabetes, osteoporosis, cancer, hepatitis C) and associated medication and/or treatment side effects on perceptions of physical attractiveness.

Many HIV-positive older adults who would benefit from face-to-face sexual risk reduction interventions live with serious comorbid health conditions that complicate travel to medical and social service appointments, have significant confidentiality concerns, and are geographically isolated from traditional risk reduction resources. As such, face-to-face interventions are an unrealistic intervention modality for many members of this group. However, risk reduction interventions delivered using distance technologies, such as regular and cellular telephones, can reach many older adults living with HIV/AIDS.

In response to the lack of age-appropriate risk reduction interventions for HIV-infected older adults who engage in high-risk sex, and the potential of telephone technology to deliver cost-effective risk reduction interventions to this group, this study tested the efficacy of 1- and 4-session telephone-administered behavioral sexual risk reduction interventions for HIV-positive adults 45-plus years of age who engage in risky sexual behaviors.

ELIGIBILITY:
Inclusion Criteria:

* HIV-positive
* English-speaking
* Access to a land line or cellular telephone
* Unprotected anal or vaginal intercourse in the past 3 months

Exclusion Criteria:

* Sexual partner of study participant

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2009-11; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Change in self-reported number of non-condom-protected anal and vaginal sex acts in the past 3 months from baseline to 3-month follow-up | baseline, 3-month follow-up
Change in self-reported number of non-condom-protected anal and vaginal sex acts in the past 3 months from baseline to 6-month follow-up | baseline, 6-month follow-up

SECONDARY OUTCOMES:
Proportion of participants reporting 100% condom use for anal and vaginal sex in the past 3 months | 3-month follow-up, 6-month follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Travis I Lovejoy, Ph.D., M.P.H., Principal Investigator — Ohio University College of Osteopathic Medicine
Locations (1):
- Ohio University College of Osteopathic Medicine, Athens, Ohio, United States

REFERENCES:
- [Result] Lovejoy TI, Heckman TG, Suhr JA, Anderson T, Heckman BD, France CR. Telephone-administered motivational interviewing reduces risky sexual behavior in HIV-positive late middle-age and older adults: a pilot randomized controlled trial. AIDS Behav. 2011 Nov;15(8):1623-34. doi: 10.1007/s10461-011-0016-x. PMID 21809048